CLINICAL TRIAL: NCT06609317
Title: Feasibility of Pelvic Floor Muscle Training With a Digital Therapeutic Motion-based Device (Leva Device) in a Postpartum Population
Brief Title: Postpartum pElvic Assisted Recovery With Leva
Acronym: PEARL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 007382
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Postpartum Pelvic Floor Function and Symptoms
Keywords: postpartum pelvic muscle training; postpartum pelvic floor; postpartum pelvic floor physical therapy; postpartum urinary incontinence; postpartum bowel incontinence; postpartum pelvic floor recovery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device Arm (Experimental): Participants in this arm will use a digital therapeutic motion-based device for postpartum pelvic floor muscle training
  Interventions: Device: Digital therapeutic motion-based device

INTERVENTIONS:
Device: Digital therapeutic motion-based device — This intervention includes use of a digital therapeutic motion-based device for pelvic floor muscle training

SUMMARY:
The goal of this prospective cohort study is to evaluate the feasibility of postpartum pelvic floor muscle training using an FDA-cleared digital therapeutic motion-based device.

In addition to assessing feasibility, investigators also will evaluate bladder and bowel function, pelvic organ prolapse symptoms, and vaginal and perineal pain in the immediate postpartum period and at 3 and 6 months postpartum. Investigators also will assess sexual function at 3 and 6 months postpartum.

Participants will use the motion-based device for postpartum pelvic floor muscle training and will complete electronically administered surveys at 3 and 6 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous vaginal delivery within the last 4-8 weeks
* Age ≥ 18 years
* Ambulatory
* Willing and able to consent to participate.
* English speaking
* Owns a smartphone

Exclusion Criteria:

* Operative or cesarean delivery
* Obstetric delivery at less than 20 weeks gestation
* Third- or fourth-degree perineal laceration
* Episiotomy
* Multiples

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-04-04 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility | From enrollment to 6 months postpartum
  Feasibility will be assessed using participant reported discomfort with device use, ease of device use, net promotor score, patient satisfaction, and free text feedback on the device.
Perineal Pain | From enrollment to 6 months postpartum
  Participants will complete validated surveys assessing perineal pain at baseline, 3 months postpartum, and 6 months postpartum.

SECONDARY OUTCOMES:
Bladder function | From enrollment to 6 months postpartum
  Participants will complete validated surveys assessing bladder function at baseline, 3 months postpartum, and 6 months postpartum.
Bowel Function | From enrollment to 6 months postpartum
  Participants will complete validated surveys assessing bowel function at baseline, 3 months postpartum, and 6 months postpartum.
Pelvic Organ Prolapse | From enrollment to 6 months postpartum
  Participants will complete validated surveys assessing pelvic organ prolapse symptoms at baseline, 3 months postpartum, and 6 months postpartum.
Vaginal pain | From enrollment to 6 months postpartum
  Participants will complete validated surveys assessing vaginal pain at baseline, 3 months postpartum, and 6 months postpartum.
Sexual function | From enrollment to 6 months postpartum
  Participants will complete validated surveys assessing sexual function at 3 months postpartum and 6 months postpartum.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of South Florida, Tampa, Florida
  - Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No